CLINICAL TRIAL: NCT04622969
Title: Targeting Behavioral Adjustment and Healthy Lifestyle in Preschool-age Children Using an Integrated Family-Based Intervention
Brief Title: The Healthy Child Development Program Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Ron Prinz, PhD, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00091502
Record Dates: First submitted 2020-10-24; First posted 2020-11-10 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Child Behavior; Child Health; Child, Preschool; Parents
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Provide the 15-week Healthy Child Development Program intervention
  Interventions: Behavioral: Healthy Child Development Program
- Wait list control (No Intervention): Not provide the Healthy Child Development Program during study:
  Individuals in this condition do not participate in the intervention program until after the study period is completed.

INTERVENTIONS:
Behavioral: Healthy Child Development Program — The Healthy Child Development Program is a family-based intervention focused on strengthening positive behaviors in children, managing misbehavior, and addressing healthy lifestyle choices.
  Arms: Intervention

SUMMARY:
This study conducts a preliminary test of an intervention program delivered in the home to assist families of preschool-age children with social, emotional, and behavioral development, and the acquisition of healthy lifestyle behaviors.

DETAILED DESCRIPTION:
Utilizing referrals from community-based organizations serving high-risk families, this study addresses both health and behavioral domains through a family-based intervention. The home-delivered prevention intervention includes content on strengthening positive behaviors in children, managing misbehavior, and addressing healthy lifestyle choices. Families engage in practical skill building and have the opportunity to practice these skills and receive feedback.

ELIGIBILITY:
Inclusion Criteria:

* parent has primary custody of the child
* one or more children in the home is in the 3 to 4 year old age range
* English-speaking parent
* parent stated an interest to participate in the program
* parent completes informed consent process
* family experiencing economic disadvantage
* parenting challenges due to child behavior

Exclusion Criteria:

* an open Child Protective Services maltreatment case on the family
* parent receiving inpatient treatment or enrolled in an institutional-residential treatment program

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen D Seay, Ph.D., MSW, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Wait List Control: Not provide the Healthy Child Development Program during study
  Individuals in this condition do not participate in the intervention program until after the study period is completed.
Period: Overall Study
Arm/Group | Intervention | Wait List Control
Started | 31 | 32
Completed | 29 | 29
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait List Control | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.03 (0.66) | 3.98 (0.79) | 4.01 (0.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Child Gender: Female | 10 | 8 | 18
  Child Gender: Male | 21 | 24 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 27 | 30 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 13 | 23
  White | 15 | 14 | 29
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63
Baseline Outcome Measure Child Behavior Problems [Mean (Standard Deviation); unit: units on a scale] | 132.8 (35.5) | 145.4 (30.9) | 139.2 (33.2)

OUTCOME MEASURES:

1. Primary Outcome: Child Behavior Problems
Description: Child behavior problems refers to the Eyberg Child Behavior Inventory Intensity Scale, which is the sum of parental report responses on 36 items. The minimum and maximum values on this measure are 36 and 252 respectively, with higher scores meaning a worse outcome.
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 132.8 (35.5) | 145.4 (30.9)

2. Primary Outcome: Child Behavior Problems
Description: as for outcome 1
Time Frame: six months after baseline assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 108.2 (31.4) | 139.1 (30.3)
Statistical Analysis 1: Comparison: Intervention vs Wait List Control; Test type: Superiority; p < .001, ANCOVA; Mean Difference (Net) = -21.60, Standard Error of Mean 5.157

3. Primary Outcome: Child Physical Activity
Description: Child physical activity will be measured using an ActiGraph Link accelerometer to assess the number of minutes each day for each level of activity, to arrive at the average number of minutes per day the child spends engaging in moderate and vigorous physical activity.
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
minutes | 91.9 (6.99) | 92.9 (6.49)

4. Primary Outcome: Child Physical Activity
Description: as for outcome 3
Time Frame: six months after baseline assessment
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
minutes | 88.6 (7.13) | 82.5 (7.40)
Statistical Analysis 1: Comparison: Intervention vs Wait List Control; Test type: Superiority; p = 0.56, Mixed Models Analysis; Mean Difference (Net) = 7.12, Standard Error of Mean 12.05

5. Primary Outcome: Child Screen Time
Description: Multi-day estimate of child screen time will be derived from parental log for the daily amount of child screen time at home.
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Error); unit: hours
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
hours | 1.59 (0.21) | 2.29 (0.21)

6. Primary Outcome: Child Screen Time
Description: as for outcome 5
Time Frame: six months after baseline assessment
Measure: Mean (Standard Error); unit: hours
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
hours | 1.35 (0.21) | 2.00 (0.21)

7. Primary Outcome: Child Sleep Duration
Description: Multi-day estimate of child sleep duration will be derived from parental log for the daily amount of child sleep duration at home.
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Error); unit: hours
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
hours | 10.4 (0.14) | 10.2 (0.14)

8. Primary Outcome: Child Sleep Duration
Description: as for outcome 7
Time Frame: six months after baseline assessment
Measure: Mean (Standard Error); unit: hours
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
hours | 10.4 (0.15) | 10.1 (0.15)
Statistical Analysis 1: Comparison: Intervention vs Wait List Control; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Net) = 0.0015, Standard Error of Mean 0.145

9. Secondary Outcome: Parenting Difficulties
Description: Parenting difficulties refers to the Parenting Scale Total Score. The total score is the average of 30 items, with a minimum value of 1.0 and a maximum value of 7.0. Higher scores mean a worse outcome (i.e., greater parenting difficulties).
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 3.29 (0.78) | 3.29 (0.65)

10. Secondary Outcome: Parenting Difficulties
Description: as for outcome 9
Time Frame: six months after baseline assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 2.90 (0.71) | 3.17 (0.63)
Statistical Analysis 1: Comparison: Intervention vs Wait List Control; Test type: Superiority; p < .05, ANCOVA; Mean Difference (Net) = -0.264, Standard Error of Mean 0.121

11. Secondary Outcome: Parental Stress
Description: Parental stress refers to the Parenting Daily Hassles Scale, which is the total of 20 items. The minimum and maximum values are 0 and 80 respectively, with higher scores meaning a worse outcome (i.e., greater parental stress).
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 47.3 (13.1) | 47.2 (7.8)

12. Secondary Outcome: Parental Stress
Description: as for outcome 11
Time Frame: six months after baseline assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 40.24 (10.5) | 45.72 (9.07)
Statistical Analysis 1: Comparison: Intervention vs Wait List Control; Test type: Superiority; p < .01, ANCOVA; Mean Difference (Net) = -5.573, Standard Error of Mean 1.802

13. Secondary Outcome: Parental Confidence
Description: Parental confidence refers to the Parenting Sense of Competence scale. This scale, based on the sum of responses on 17 items, ranges from a minimum of 17 and a maximum of 102, with higher scores meaning a better outcome (i.e., greater parental confidence).
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 68.3 (10.7) | 71.6 (9.7)

14. Secondary Outcome: Parental Confidence
Description: as for outcome 13
Time Frame: six months after baseline assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 31 | 32
score on a scale | 74.96 (10.48) | 73.79 (9.40)
Statistical Analysis 1: Comparison: Intervention vs Wait List Control; Test type: Superiority; p = .062, ANCOVA; Mean Difference (Net) = 3.509, Standard Error of Mean 1.842
Statistical Analysis 2: Comparison: Intervention vs Wait List Control; Test type: Superiority; p = 0.78, Mixed Models Analysis; Mean Difference (Net) = 0.047, Standard Error of Mean 0.170

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT04622969/Prot_SAP_000.pdf